CLINICAL TRIAL: NCT06624111
Title: Assessing Weight Bias Among Turkish Dietitians: Determinants and Impact on Professional Practice
Brief Title: Assessing Weight Bias Among Turkish Dietitians
Status: Completed | Type: Observational
Sponsor: Ezgi Bellikci Koyu (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ezgi Bellikci Koyu, Assistant Professor, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Other Study IDs: 1919B012005303
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Weight Bias; Weight Stigma
Keywords: obesity; weight bias; weight stigma; fat-phobia; dietitian
MeSH Terms: conditions — Weight Prejudice; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Picture belong to a patient with obesity: Dietitians were randomly assigned to a case study via SurveyMonkey. All the information (demographics, biochemical parameters and diet history physical activity level) about the cases was the same, only their weight and, therefore, their photographs were different. In this case there was a photograph of a woman with obesity
- Picture belong to a patient with normal-weight: Dietitians were randomly assigned to a case study via SurveyMonkey. All the information (demographics, biochemical parameters and diet history physical activity level) about the cases was the same, only their weight and, therefore, their photographs were different. In this case there was a photograph of a woman with normal weight.

SUMMARY:
The objective of this study was to examine weight bias among Turkish dietitians. and to investigate the effect of the patient's weight status on the dietitian's assessment and dietetic practice.

DETAILED DESCRIPTION:
The dietitians were randomly assigned to an online case study with lactose intolerance, with all patient information identical except for the patient's weight and photograph. In one case there was a photograph of a woman with obesity and in the other a woman of normal weight. The objective of the case study was to evaluate how the body weight of a patient who consulted a dietitian for a reason unrelated to the body weight affected professional practices.

ELIGIBILITY:
Inclusion Criteria:

* Dietitians working in Turkiye

Exclusion Criteria:

* Pregnancy
* breastfeeding

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study sample consisted of dietitians working Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Differences between dietitians' lifestyle recommendations among groups. | Baseline
  Dietitians' recommendations lifestyle recommendations (such as dietary intake of energy and macronutrients) were assessed using a 5-point Likert-type scale (1; should be greatly reduced, 5; should be greatly increased).

SECONDARY OUTCOMES:
Differences between the biochemical status rated by dietitians between groups | Baseline
  Dietitians rated the biochemical status of the case with a 5-point Likert type scale (1; very good, 5; very poor).
Differences between the diet quality rated by dietitians between groups | Baseline
  Dietitians rated the diet quality of the case with a 5-point Likert type scale (1; very good, 5; very poor).
Differences between dietatians' expectations regarding the patient's adherence to the diet between groups | Baseline
  Dietatians' expectations regarding the patient's adherence to the diet were assessed using the statements "the patient is willing to be treated", "the patient is expected to comply with the treatment recommendations", "the patient will be successful in making dietary changes", "the patient will be able to sustain recommendations", "the patient understood treatment recommendations". A 5-point Likert type scale (1; strongly disagree, 5; strongly agree) was used to rate these statements.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication

REFERENCES:
- [Derived] Bellikci-Koyu E, Karaagac Y, Demirci S. Assessing weight bias among Turkish dietitians: determinants and impact on professional practice. BMC Med Educ. 2025 Feb 25;25(1):307. doi: 10.1186/s12909-025-06883-8. PMID 40001117